CLINICAL TRIAL: NCT04582071
Title: Assessing Efficacy of Psychotherapy Intervention With Inflammatory Bowel Disease Surgery Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: After further review and discussion, the scope of the study is being changed to better suit the patient population. No subjects were enrolled in the study.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-00275
Record Dates: First submitted 2020-10-05; First posted 2020-10-09 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Anxiety Depression
MeSH Terms: interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Psychotherapy, Intervention arm) (Experimental): Subjects undergoing a 3 step IPAA will receive the four sessions of psychotherapy preceding and following their first surgery only, and receive an additional set of questionnaires again after their third surgery.
  Interventions: Behavioral: Psychotherapy
- Arm 2 (Non-Therapy, Control Arm) (No Intervention): Subjects will receive questionnaires which will be administered remotely via telemedicine if patient and psychologist/ research team member are unable to meet in person.

INTERVENTIONS:
Behavioral: Psychotherapy — Psychotherapy is a term that we use to describe the use of the psychological method to understand and improve an individual's well-being and mental health. The Principal Investigator of this study, a clinical psychologist will be leading each of the sessions.
  Arms: Arm 1 (Psychotherapy, Intervention arm)

SUMMARY:
The purpose of this research study is to understand the effects of therapy in lowering anxiety and improving quality of life in patients with IBD who are undergoing surgery

DETAILED DESCRIPTION:
Pre- and post- surgery scores on the State Trait Anxiety Inventory will be used to measure levels of state-based anxiety as the primary outcome. Our hypothesis is that patients in the experimental group, will show a decrease in anxiety levels over the course of the four sessions, while the same group in the control group will not change significantly in their anxiety levels. It is hypothesized that this would be due to the psychotherapeutic intervention mitigating the inherent emotional stress and negative behavioral changes associated with surgery. It will be important to differentiate between the inpatient and outpatient groups, as their anxiety levels may inherently be discrepant. For patients with a three-step ileal pouch-anal anastomosis (IPAA), the three sessions subsequent to surgery will be conducted only after the first surgery. This is an exploratory study in which we are investigating the possibility of a range of potential outcomes to the intervention, including overall reduction of anxiety, depression, body image and improvement in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients age18 years or older.
* Patients with documented diagnosis of Inflammatory Bowel Disease.
* Patients with documented need for IBD surgery

Exclusion Criteria:

* Patients younger than 18 years of age.
* Patient who has any condition, including physical, psychological, or psychiatric condition, which in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data and renders the patient an unsuitable candidate for the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change in State - based anxiety | Visit 1 (2 Weeks Pre-Surgery Visit), Visit 4 (3 months after surgery) Visit 5 (Approximately 6 months post-administration of last session)
  State based anxiety will be measured by the State-Trait Anxiety Inventory. This measure has 40 items. Range of scores for each subtest is 20-80, the higher score indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms for the S-Anxiety scale.

SECONDARY OUTCOMES:
Change in participant's level of depression | Visit 1 (2 Weeks Pre-Surgery Visit), Visit 4 (3 months after surgery) Visit 5 (Approximately 6 months post-administration of last session)
  Measured by PHQ-9- Patient Health Questionnaire. Questionnaire has 9 items scores each of the nine DSM-IV criteria as "0" (not at all) to "3". Subjects will achieve one out of four levels of depression severity, depending upon their scores: 0-4=minimal or none, 5-9=mild, 10-14=moderate, and 15-19=moderately severe to severe.
Change in Quality of life of participants | Visit 1 (2 Weeks Pre-Surgery Visit), Visit 4 (3 months after surgery) Visit 5 (Approximately 6 months post-administration of last session)
  Measured by IBD QoL- Inflammatory Bowel Disease Quality of Life Questionnaire. Questionnaire has 32 items and the higher scores indicate better quality of life.
Increase ability to function | Visit 1 (2 Weeks Pre-Surgery Visit), Visit 4 (3 months after surgery) Visit 5 (Approximately 6 months post-administration of last session)
  Measured by Work Productivity and Activity Impairment (WPAI). There is 6 items which yeilds four types of scores: Absenteeism (work time missed), Presenteesism (impairment at work / reduced on-the-job effectiveness), Work productivity loss (overall work impairment/absenteeism plus presenteeism) and Activity Impairment The sum of specific health problem impairment and impairment due to other health reasons is equal to impairment due to all health reasons. WPAI outcomes are expressed as impairment percentages, multiply scores by 100 to express in percentages, with higher numbers indicating greater impairment and less productivity
Improved self efficacy in participants | Visit 1 (2 Weeks Pre-Surgery Visit), Visit 4 (3 months after surgery) Visit 5 (Approximately 6 months post-administration of last session)
  Measured by The Self-Efficacy Scale with 8 items with higher scores which will indicate greater self-efficacy.
Change in social support of participants | Visit 1 (2 Weeks Pre-Surgery Visit), Visit 4 (3 months after surgery) Visit 5 (Approximately 6 months post-administration of last session)
  This will be measured by Social Support Survey which has 19 items to obtain a score for each of four subscales, calculate the average of the scores for each item in the subscale. Higher scores for an individual scale or for the overall support index indicate more support.
Improvement in coping strategies | Visit 1 (2 Weeks Pre-Surgery Visit), Visit 4 (3 months after surgery) Visit 5 (Approximately 6 months post-administration of last session)
  Measured by The Brief Cope questionnaire with 28 items which are 14 subscales with 2 items each. Sum of each subscale indicates a preference for particular coping strategies, which can be characterized as either effective or less effective.
Change in the participants perception of body image | Visit 1 (2 Weeks Pre-Surgery Visit), Visit 4 (3 months after surgery) Visit 5 (Approximately 6 months post-administration of last session)
  Measured by The Body Image Scale which includes 9 items. Participants score from 0 ("not at all") to 3 ("very much") on each of the 9 questions so that the lowest possible total score is 0 and the highest 27, with higher scores indicating increasing body image dissatisfaction.
Change in the participants' perception of illness | Visit 1 (2 Weeks Pre-Surgery Visit), Visit 4 (3 months after surgery) Visit 5 (Approximately 6 months post-administration of last session)
  Measured by The Brief Illness Perception Questionnaire which 9 items. Five of the items assess cognitive illness representations: consequences (Item 1), timeline (Item 2), personal control (Item 3), treatment control (Item 4), and identity (Item 5). Two of the items assess emotional representations: concern (Item 6) and emotions (Item 8). One item assesses illness comprehensibility (Item 7). Assessment of the causal representation is by an open-ended response item adapted from the IPQ-R, which asks patients to list the three most important usual factors in their illness (Item 9). Responses to the causal item can be grouped into categories such as stress, lifestyle, hereditary, etc., determined by the particular illness studied, and categorical analysis can then be performed.
  The Brief IPQ allows very simple interpretation of scores: increases in item scores represent linear increases in the dimension measured.
Change in pain perception | Visit 1 (2 Weeks Pre-Surgery Visit), Visit 4 (3 months after surgery) Visit 5 (Approximately 6 months post-administration of last session)
  Measured by Pain anxiety symptom scale short form 20 with 20 items. The PASS assesses pain-specific anxiety symptoms and consists of four 10-item subscales measuring cognitive anxiety responses, escape and avoidance, fearful thinking and physiological anxiety responses. Higher scores indicate greater anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Gerson, MD, Principal Investigator — NYU Langone Health

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to Ghoncheh.Ghiasian@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.